CLINICAL TRIAL: NCT01609413
Title: A Human Crossover Study to Compare the Bioavailability of Calcium From AlgaeCal® Versus a Proprietary Calcium Dietary Supplement
Brief Title: The COMparison of CALcium Bioavailability Between AlgaeCal® and a Proprietary Supplement
Acronym: COMCAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sprim Italia (Unknown)
Collaborators: AlgaeCal Inc. (Industry)
Responsible Party: Sponsor
Organization: SPRIM Advanced Life Sciences, SprimItalia (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: #09-MAX-05-BIO-01b; NCT01022593 (obsolete NCT alias)
Record Dates: First submitted 2012-05-23; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AlgaeCal (Experimental): Calcium supplements derived from ocean algae. One dose equals 3 capsules containing 180 mg calcium each.
  Interventions: Dietary Supplement: AlgaeCal
- Caltrate 600 (Active Comparator): Proprietary calcium supplement. One dose contains 600 mg of calcium.
  Interventions: Dietary Supplement: Caltrate 600

INTERVENTIONS:
Dietary Supplement: AlgaeCal — One dose equals 3 times 180 mg of calcium, to be taken one time on the morning of the examination day.
  Arms: AlgaeCal
Dietary Supplement: Caltrate 600 — One dose equals 1 capsule of 600 mg calcium, to be taken one time on the morning of the examination day.
  Arms: Caltrate 600

SUMMARY:
In a crossover, single blind, randomized trial the calcium bioavailability of two calcium supplements will be compared.That is AlgaeCal®(Algaecal Inc, Vancouver, Canada)(1 dose is 3 capsules of 180 mg calcium), derived from ocean algae and the proprietary calcium supplement Caltrate 600® (Wyeth Consumer Healthcare, Inc).

After a screening visits 20 healthy male subjects aged 20-50 years will spend a day at the research center to examine calcium bioavailability data. They will be randomized to consume either first the AlgaeCal® supplement or the Caltrate 600® supplement. After a one week wash-out period subjects will be supplemented with the other supplement. During the examination day blood and urine samples will be collected before and until eight hours after the supplementation for analyses of calcium, creatinine, phosphorus, albumin and 25 Hydroxy vitamin D. Subjects are instructed to avoid taking calcium and/or vitamin D supplements 1 week before and during the entire study period. In addition, they are not allowed to take medication that may affect calcium metabolism.

The hypothesis of the study is that calcium bioavailability of the AlgaeCal® supplement will be higher than that of the Caltrate 600® supplement.

DETAILED DESCRIPTION:
This was a single centre, single-dose, randomized, two way cross-over study in healthy male subjects.

The study consisted of the following visits:

1. A screening visit to select eligible subjects according to the inclusion/exclusion criteria detailed in the study protocol.
2. Visit 1 in which subjects who satisfied the selection criteria were assigned to one of the two intervention sequences (Algaecal®/ LCCS or LCCS/Algaecal®) according to the randomization list;
3. Visit 2, after at least one week of wash-out in respect to visit 1. Subjects arrived at the centre early in the morning The first blood sample was drawn before the ingestion of the calcium supplement and every hour after for the following 8 hours. Urine sample were collected before the ingestion of the calcium supplement and every 2 hours after for the following 8 hours. During each study visit the subjects were present in the site centre from the morning to the evening. Calcium supplement was given under fasted condition and during the eight hours after the product ingestion, according to the protocol, only water ad libitum was allowed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living men aged 20 to 50 years-old
* Consent to the study and compliance with study product

Exclusion Criteria:

* Calcium supplements or calcitriol taken one week or less before the first kinetic visit
* Heart disease
* Circulation problems
* Parathyroid gland disorder
* Kidney disease
* Past or present kidney stones
* Gastrointestinal disturbances that could potentially affect the absorption of calcium supplements

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Will be measured the oral bioavailability of calcium from a single dose of AlgaeCal® (Algaecal, Vancouver, Canada) compared to a proprietary calcium supplement (Caltrate 600®, Whyett Consumer healthcare, Inc). | one day
  During the examination day blood and urine samples will be collected before and untill eight hours after the supplementation for analyses of calcium, creatinine, phosphorus, albumin and 25 Hydroxy vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Clementi, Prof, Principal Investigator — University of Milan, Milan, Italy
Locations (1):
- Luigi Sacco Hospital, Milan, Milan, Italy